CLINICAL TRIAL: NCT03380936
Title: A Randomized Pilot Study of Treatment for Subclinical Antibody-Mediated Rejection in Kidney Transplant Recipients
Brief Title: Pilot Study of Treatment for Subclinical AMR (Antibody-mediated Rejection) in Kidney Transplant Recipients
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Slower than expected recruitment rate
Sponsor: University of Colorado, Denver (Other)
Collaborators: Veloxis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-1812
Record Dates: First submitted 2017-10-26; First posted 2017-12-21 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Kidney Transplant Rejection
Keywords: subclinical; graft rejection; AMR (antibody-mediated rejection); AMBR (acute antibody-mediated rejection); DSA (donor specific antibodies)
MeSH Terms: interventions — Tacrolimus; Plasma Exchange; Immunoglobulins, Intravenous

STUDY DESIGN:
Intervention Model Description: Only patients meeting histologic criteria for AMR by Banff 2013 criteria will be randomized (ptc + g + c4d ≥ 2). Subjects will be randomized to either undergo optimization (conversion to Envarsus with goal trough tacrolimus level > 8 ng/ml, mycophenolic acid at 720 mg, prednisone at current dose (5mg) or continue taper to 5mg per center standard of care protocol of or treatment.); or, to treat clinical AMR (antibody mediated rejection) with plasma exchange x 5 treatments, each followed by IVIG (intravenous immunoglobulin) 200 mg/kg except last dose of 1 gm/kg. Rituximab 375 mg/m2 following final plasma exchange treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 - conversion to Envarsus XR (Active Comparator): Optimize: conversion to Envarsus XR (Tacrolimus Extended Release Oral Tablet [Envarsus]) with goal trough tac level > 8 ng/ml, MPA at 720 mg bid unless medically contraindicated, prednisone at current dose (5mg) or continue taper to 5mg per center standard of care protocol
  Interventions: Drug: Tacrolimus Extended Release Oral Tablet [Envarsus]
- Arm 2 - plasma exchange and IVIG (Active Comparator): Treat clinical AMR: Plasma exchange x 5 treatments, each followed by IVIG 200 mg/kg except last dose of 1 gm/kg. Rituximab 375 mg/m2 following final plasma exchange treatment.
  Interventions: Other: Plasma Exchange and IVIG (Intravenous Immunoglobulin )

INTERVENTIONS:
Drug: Tacrolimus Extended Release Oral Tablet [Envarsus] — Switching from current version of tacrolimus to the extended release, once a day version (Envarsus) and titrating dose to achieve an optimal trough level. Goal trough tac level > 8 ng/ml, MPA at 720 mg bid unless medically contraindicated, prednisone at current dose (5mg) or continue taper to 5mg per center standard of care protocol.
  Other Names: Envarsus XR
  Arms: Arm 1 - conversion to Envarsus XR
Other: Plasma Exchange and IVIG (Intravenous Immunoglobulin ) — Plasma exchange x 5 treatments, each followed by IVIG 200 mg/kg except last dose of 1 gm/kg. Rituximab 375 mg/m2 following final plasma exchange treatment.
  Arms: Arm 2 - plasma exchange and IVIG

SUMMARY:
This is a pilot study to determine if extended release Envarsus at an optimal level is just as effective as more invasive standard therapies for subclinical (mild) AMR (antibody mediated rejection) in kidney transplant patients. Subjects will be randomized to either conversion to Envarsus XR (extended release); or, to a standard of care regimen of plasma exchange/IVIG (intravenous immunoglobulin)/rituximab treatments.

DETAILED DESCRIPTION:
There is currently minimal data to guide treatment of mild graft damage in kidney transplant patients. Some of the current therapies used often come with dangerous complications (infections, malignancies, etc.). This is a pilot study to determine if extended release Envarsus at an optimal level is just as effective as more invasive standard therapies for subclinical (mild) AMR (antibody mediated rejection) in kidney transplant patients. The subjects will be randomized to either conversion from their current tacrolimus regimen to Envarsus XR (a once a day, extended release version of tacrolimus); or, to a regimen of 5 plasma exchanges/IVIG (intravenous immunoglobulin) treatments and one treatment with rituximab. Subjects who are within their first year of transplant will visit their doctor monthly for regular tests and checks and then will have a kidney biopsy at 6 months. Subjects who had their transplant over a year prior will see the doctor for tests and checks at 1, 3 and 5 months and then will have a biopsy of the kidney at month 6.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18+ years) recipients of kidney or kidney/pancreas transplants
* Willing to sign an IRB (institutional review board)-approved consent and to comply with study requirements
* DSA (donor specific antibodies) detected by SAB (single antigen beads) screening with MFI ≥ 2000
* Graft biopsy performed within prior 30 days
* Stable renal function defined by serum creatinine increase ≤ 30% over prior 6 months
* Subacute antibody-mediated rejection on biopsy defined by ptc + g + C4d ≥ 2 by Banff 2013 criteria

Exclusion Criteria:

* Kidney/liver or kidney/heart recipient
* Unwilling/unable to undergo screening biopsy
* HIV (human immunodeficiency virus), HCV (hepatitis-C virus), or HBsAg (hepatitis-B surface antigen) positive
* Active/untreated infection
* Acute cellular rejection with Banff grade 1b, 2a, 2b on initial biopsy requiring rATG (rabbit anti-thymocyte globulin) therapy
* Pregnant or nursing females

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-01-17 (Actual); Primary Completion 2019-10-16 (Actual); Study Completion 2019-10-16 (Actual)

PRIMARY OUTCOMES:
Change in Acute Inflammatory Histologic Parameters | Baseline and 6 months
  Any increase or reduction in ptc+g+C4d score by Banff 2013 criteria) from baseline (pre-treatment) to 6 month (post-treatment initiation). Analysis will comprise exact chi-squared tests for comparison of binomial proportions of histological response between the two treatment groups.

SECONDARY OUTCOMES:
Change in MDRD GFR (Modification of Diet in Renal Disease Glomerular Filtration Rate) | 6 and 12 months
  Comparison of these levels and any changes of levels/rates using two-sided two-sample t-tests.
Change in Donor-Specific Antibody (DSA) Mean Fluorescence Intensity (MFI) Level | 6 and 12 months
  Comparison of these levels and any changes of levels/rates using two-sided two-sample t-tests.
Change in serum creatinine | 6 and 12 months
  Comparison of these levels and any changes of levels/rates using two-sided two-sample t-tests.
Graft Survival | 6 and 12 months
  Total and death-censored calculated using Kaplan-Meier methods and compared using logrank tests.
Patient Survival | 6 and 12 months
  Total and death-censored calculated using Kaplan-Meier methods and compared using logrank tests.
Evaluation of Adverse Events | 6 and 12 months
  All potential adverse events will be captured and recorded by study coordinators during post-treatment standard of care clinic visits, and reviewed by PI. Adverse events will be reported for each group separately and compared using exact chi-squared tests.

CONTACTS AND LOCATIONS:
Overall Officials: James Cooper, M.D., Principal Investigator — University of Colorado, Denver; Scott Davis, M.D., Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No